CLINICAL TRIAL: NCT07222163
Title: Stuttering and Neuromodulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25-00866
Record Dates: First submitted 2025-10-28; First posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Stuttering
Keywords: tDCS
MeSH Terms: conditions — Stuttering

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Behavioral speech therapy combined with active tDCS (Experimental): Each participant will complete ten treatment sessions over approximately ten weeks. In each session, participants will receive active tDCS for 30 minutes while concurrently engaging in behavioral speech therapy. Active stimulation will include a 30-second ramp-up to 2.0 mA, 30 minutes of continuous stimulation, and a 30-second ramp-down.
  Interventions: Device: Soterix Medical 1x1 tDCS system; Behavioral: Speech therapy sessions
- Behavioral speech therapy combined with sham tDCS (Sham Comparator): Each participant will complete ten treatment sessions over approximately ten weeks. In each session, participants will receive sham tDCS for 30 minutes while concurrently engaging in behavioral speech therapy. Sham stimulation will involve the same ramp-up and ramp-down but with no current delivered during the 30-minute period to maintain blinding.
  Interventions: Device: Soterix Medical 1x1 tDCS system; Behavioral: Speech therapy sessions

INTERVENTIONS:
Device: Soterix Medical 1x1 tDCS system — Stimulation (2.0 mA for 30 minutes) will occur during speech therapy sessions focused on practicing speech techniques. Sham stimulation will mimic the physical sensation without active current.
Behavioral: Speech therapy sessions — Each of the ten weekly sessions will begin with 15 minutes of strategy practice, providing participants with the opportunity to rehearse light contact and easy onset techniques prior to the tDCS-enhanced speaking task.

SUMMARY:
The purpose of this study is to collect preliminary data on the efficacy of transcranial direct current stimulation (tDCS) combined with traditional behavioral techniques to reduce stuttering severity and negative impact in adults who stutter. The study also aims to explore neuroplastic changes (i.e., regional activation and functional connectivity) resulting from combined tDCS + speech therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 to 65 years.
2. Diagnosis of developmental stuttering, verified by a licensed speech-language pathologist.
3. Mild-to-moderate or greater stuttering severity, defined as a score of 20 or higher on the Stuttering Severity Instrument-Fourth Edition (SSI-4).
4. English as a primary language.
5. Right-handedness (to minimize variability in neural lateralization).
6. Willing and able to attend all study sessions and follow study procedures.

Exclusion Criteria:

1. Have a history of neurological, psychiatric, or medical conditions that are contraindicated for tDCS.
2. Are currently taking medications known to affect cortical excitability.
3. Have a history of seizures or epilepsy.
4. Are pregnant or planning to become pregnant during the study period.
5. Have metal implants in the head (excluding dental work) or other contraindications to electrical brain stimulation.
6. Any skin disorder or skin sensitive area near stimulation locations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Change in Stuttering Severity Instrument - 4th Edition (SSI-4) total score | Baseline, Visit 15 (~1-2 weeks post-intervention)
  The Stuttering Severity Instrument-4th Edition (SSI-4) provides a total score that is compared to age-specific norms to determine severity, with ranges for "Very Mild" to "Very Severe". The SSI-4 calculates individual scores for frequency (2-18), duration (2-18), and physical concomitants (0-20). These individual scores are combined to create a total score, which is then ranked against norms to provide a verbal severity descriptor, such as mild, moderate, severe, or very severe.
Change in the Wright and Ayre Stuttering Self-Rating Profile (WASSP) score | Baseline, Visit 15 (~1-2 weeks post-intervention)
  The WASSP produces a profile of scores across five subscales. There is a total of 26 items each scored on a seven-point Likert-type scale. A score of '1' represents the least severe/negative perception, while a '7' represents the most severe/negative perception on each scale. Total scores range from 26-182, with higher scores indicating a greater negative impact of stuttering on their life.
Stuttering impact as assessed by the Overall Assessment of the Speaker's Experience of Stuttering - Adults (OASES-A) | Baseline, Visit 15 (~1-2 weeks post-intervention)
  The OASES-A is a tool used by speech-language pathologists to measure the adverse impact of stuttering on an adult's life. It consists of 100 questions rated on a 5-point scale (1-5). The scores from individual questions are added together to create an overall score. The total score is then used to determine the "Impact Rating" on a scale from mild to severe. Higher scores indicate higher levels of negative impact.
Change in the Brief Version of the Unhelpful Thoughts and Beliefs About Stuttering Scales (UTBAS-6) total score | Baseline, Visit 15 (~1-2 weeks post-intervention)
  The UTBAS-6 is a six-item screening questionnaire for adults who stutter to measure unhelpful thoughts and beliefs associated with speech anxiety. The UTBAS-6 has a subscale score range of 6 to 30 and a total score range of 18 to 90. A higher score indicates more frequent unhelpful thoughts and greater anxiety related to stuttering.
Change in Brief Fear of Negative Evaluation (BFNE-S) Scale total score | Baseline, Visit 15 (~1-2 weeks post-intervention)
  The BFNE-S consists of 8 items that are rated on a five-point likert scale from 1 (not at all characteristic) to 4 (extremely characteristic). Scores range from 0 to 32. A score of 25 or higher may indicate clinically significant social anxiety.
Social Interaction Anxiety Scale (SIAS) | Baseline, Visit 15 (~1-2 weeks post-intervention)
  The SIAS is a 20-item self-report questionnaire that measures the severity of social anxiety. Each item is rated from 0 (not at all characteristic or true of me) to 4 (extremely characteristic or ture of me). Scores can range from 0 (no social anxiety) to 80 (maximum social anxiety). A score of 36 or higher is often considered clinically significant, suggesting the presence of social anxiety.

SECONDARY OUTCOMES:
Change in regional activation in/between cognitive control and speech motor areas during a delayed-naming task | Baseline, Visit 15 (~1-2 weeks post-intervention)
  Neuroplastic changes will be assessed using functional near-infrared spectroscopy (fNIRS) to measure cortical activation patterns (i.e., regional activation, functional connectivity) in/between cognitive control and speech motor areas during a delayed-naming task (pre- and post-intervention).
Change in functional connectivity in/between cognitive control and speech motor areas during a delayed-naming task | Baseline, Visit 15 (~1-2 weeks post-intervention)
  Neuroplastic changes will be assessed using functional near-infrared spectroscopy (fNIRS) to measure cortical activation patterns (i.e., regional activation, functional connectivity) in/between cognitive control and speech motor areas during a delayed-naming task (pre- and post-intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Eric S. Jackson, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting researcher provide a methodologically sound proposal and executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: Ej34@nyu.edu. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Researchers who provide a methodologically sound proposal will be granted access upon reasonable request. Requests should be directed to Ej34@nyu.edu. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.